CLINICAL TRIAL: NCT02711592
Title: Utilizing Pharmacogenomics Information in Enhancing Post-operative Total Joint Replacement Pain Management: A Pilot Study
Brief Title: Pharmacogenomics Information in Enhancing Post-operative Total Joint Replacement Pain Management: a Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-037
Record Dates: First submitted 2016-03-13; First posted 2016-03-17 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2018-10

CONDITIONS: Arthroplasty, Replacement, Knee; Pain, Postoperative
Keywords: Orthopaedic Pain Management
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genetic Panel for Analgesics (Other): Genetic testing for analgesics prior to surgery will be conducted. The subject will receive postoperative analgesia based on test results.
  Interventions: Genetic: Genetic Panel for Analgesics

INTERVENTIONS:
Genetic: Genetic Panel for Analgesics — All patients will receive genetic test panel to determine individualized optimal pain management following Total Knee Arthroplasty.

SUMMARY:
The objective of this study is to see how pain management and its outcomes are effected when pharmacogenomic testing is used to determine patient specific pain medication and dosing. Our goal is to determine if through the use of analgesic genetic testing, TKA post-operative patients will see a decrease in narcotic consumption, postsurgical opioid- related adverse reactions, and length of stay, overall NRS pain scores and while maintaining or improving their satisfaction scores.

DETAILED DESCRIPTION:
This is a pilot study that will look at how pain management will be effected when pharmacogenomic testing is utilized to select and dose narcotic pain medications prescribed for breakthrough pain in post-operative total knee arthroplasty (TKA) patients. Patients will receive individualized analgesics and doses for pain mitigation based on genetic testing results. Post op pain scores, narcotic consumption, adverse reactions, length of stay and patient satisfaction with pain management will be collected and analyzed to determine the significance of the pharmacogenomic analgesic testing.

Due to the lack of literature and evidence surrounding pharmacogenomics and its use in selecting analgesics to control post-operative pain a pilot study is being conducted to evaluate effect size (statistical variability) in an attempt to predict an appropriate sample size for a larger scale randomized control trial. The subjects enrolled and data collected for this internal pilot will be used in the larger scale parent study as well.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing total knee arthroplasty Patients able to understand study intent, and agree to study participation. Patients with a history of preoperative narcotic dependence and/or, adverse reactions to narcotics, and/or have experienced ineffective pain management with narcotics.

Exclusion Criteria:

Patients with orthopaedic and medical co-morbidities that would thwart postoperative pain control such as extra-articular pathology with referred pain to the knee (spinal stenosis, neuropathy,ipsilateral hip disease), severe knee deformity, post-traumatic and inflammatory arthritis Patients with chronic pain disorders BMI > 40 ASA class > III GI bleed within 6 months of surgery History of drug or alcohol abuse Patients unable to receive multimodal pain remitting agents including Celecoxib and Pregabalin.

Patients with diabetes and patients who are unable to receive decadron Any patient receiving general anesthesia Patients who will need to go to an ECF upon discharge Patients who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Pain Scores | Surgery to 6 weeks postop (+/- 2 weeks)
  Numerical patient reported pain scales.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Snyder, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No